CLINICAL TRIAL: NCT05456620
Title: Effectiveness of Reducing Tendon Compression in the Treatment of Insertional Achilles Tendinopathy: a Randomised Clinical Trial
Brief Title: Effectiveness of Reducing Tendon Compression in the Treatment of Insertional Achilles Tendinopathy
Acronym: GhenTendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-11818
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Insertional Achilles Tendinopathy
Keywords: Exercise therapy; Tendon compression; Tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator (LP) will be blinded to the assigned treatment throughout the data collection period. During the study, patients will be asked not to discuss their treatment exercises with the principal investigator but to consult an independent second sports physician (AB) if they have any questions about the therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Tendon Compression Rehabilitation (LTCR) (Experimental): A progressive, criteria-based, 4-stage exercise protocol in which the amount of tendon compression is limited (12 weeks).
  Interventions: Other: Exercise therapy
- High Tendon Compression Rehabilitation (HTCR) (Active Comparator): A progressive, criteria-based, 4-stage exercise protocol in which the amount of tendon compression is not limited (12 weeks).
  Interventions: Other: Exercise therapy (usual care)

INTERVENTIONS:
Other: Exercise therapy — The intervention treatment consists of a progressive 4-stage, criteria-based exercise protocol, in which the amount of tendon compression is limited. This includes:
  1. Education: Specific information on the importance of limiting tendon compression during rehabilitation, as well as general information on load management, the importance of active exercise therapy and setting expectations.
  2. Orthotic treatment: heel inserts to reduce ankle dorsiflexion during daily activities and sports
  3. Physiotherapy: Progressive tendon-loading exercise therapy (4 phases) restricting the amount of tendon compression by limiting dorsiflexion of the ankle and prohibiting stretching
  Arms: Low Tendon Compression Rehabilitation (LTCR)
Other: Exercise therapy (usual care) — The control treatment consists of a progressive 4-phase, criteria-based exercise protocol, in which the amount of tendon compression is not limited. This includes:
  1. Education: general information on load management, the importance of active exercise therapy and setting expectations.
  2. No orthotic treatment.
  3. Physiotherapy: Progressive tendon-loading exercise therapy (4 phases) without any restriction around tendon compression and encouraging stretching
  Arms: High Tendon Compression Rehabilitation (HTCR)

SUMMARY:
Insertional Achilles tendinopathy is a disabling injury that is common in running athletes. Exercise therapy is considered the best treatment option, but there is still no agreement on the modalities. For example, it is thought that compression overload may be a major cause of tendinopathy and should therefore be restricted during rehabilitation. However, this recommendation is based on expert opinion and not on hard scientific evidence. Therefore, this randomised controlled trial (RCT) will investigate whether a therapy that limits the amount of compression of the tendon during a progressive tendon-loading rehabilitation protocol actually has better outcomes in athletes with insertional Achilles tendinopathy.

Athletes with insertional Achilles tendinopathy will be randomised into two treatment groups; (1) an experimental rehabilitation protocol in which the amount of tendon compression is limited and (2) a control rehabilitation protocol in which the amount of tendon compression is not limited and is rather high. Both treatments consist of supervised progressive tendon-loading exercise therapy and patient education. In addition, the experimental group will also receive heel inserts to limit the amount of dorsiflexion during sports or daily activities. At baseline, at 12 weeks (end of intervention) and at 24 weeks (follow-up), pain, functionality, structure and intratendinous pressure will be determined.

DETAILED DESCRIPTION:
Achilles tendinopathy is a debilitating injury that is common among athletes, especially those involved in running sports. Around 30% of all runners exhibit Achilles tendinopathy with an annual incidence of 7-9%. Of these patients, roughly one-third will have insertional Achilles tendinopathy (IAT). Several mechanisms are considered to play a role in the aetiology of Achilles tendinopathy, yet a prominent role seems present for excessive overload. Traditionally, the nature of this overload is thought to be purely tensile. However, the Achilles tendon can also be exposed to compressive loads at the insertion when the tendon wraps around the posterior prominence of the calcaneus during dorsiflexion of the ankle. The formation of fibrocartilage-like tissue, which is typically found in histological examination of tendinopathy, can be considered as an adaptation to this compressive load, driven by the tenocyte's mechanotransduction process. Therefore, it is recommended to reduce the amount of compressive load on the tendon during rehabilitation while exerting sufficient tensile load. However, these recommendations are mainly based on a pilot study and expert opinion. Therefore, this RCT investigates whether a therapy in which the amount of tendon compression is restricted during a progressive tendon-loading rehabilitation protocol actually has better outcomes in terms of pain scores, functionality and structure of the Achilles tendon in athletes with insertional Achilles tendinopathy. Limiting the amount of tendon compression on the Achilles tendon insertion will be achieved by (1) patient education, (2) heel inserts and (3) an adapted exercise regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Diagnosed with insertional Achilles Tendinopathy by a sports medicine physician
* Have experienced symptoms for more than 3 months but less than 3 years
* A severity level of less than 80 points on the VISA-A score
* Playing running-based sports at least twice a week
* Able to comply with both exercise programs

Exclusion Criteria:

* Have a history of Achilles tendon rupture or surgery
* Have other disorders of the Achilles tendon or ankle (mid-portional Achilles tendinopathy, paratenonitis, osteoarthritis,...)
* Have rheumatological disorder (e.g. Spondylitis Ankylosis)
* Have metabolic or endocrine disorders, such as type I or type II diabetes
* Have had an Achilles injection in the past 3 months
* Have other conditions that prevent following an active exercise programme
* Have already been treated with physiotherapy, shockwave therapy or orthotics in the past 3 months
* Medication use with (fluoro)quinolones antibiotic in the past 2 years
* Currently pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The change of the Victorian Institute of Sports Assessment-Achilles Questionnaire (VISA-A) score over 12 weeks | 12 weeks (at the end of intervention)
  The VISA-A score is a measure of pain and lower limb function (disability) associated with Achilles tendinopathy. A higher score indicates a better outcome and a 10 point increase is accepted as being clinically meaningful.
The change of the Victorian Institute of Sports Assessment-Achilles Questionnaire (VISA-A) score over 24 weeks | 24 weeks (at follow-up)
  The VISA-A score is a measure of pain and lower limb function (disability) associated with Achilles tendinopathy. A higher score indicates a better outcome and a 10 point increase is accepted as being clinically meaningful.

SECONDARY OUTCOMES:
Subjective patient satisfaction | This will be assessed at the end of the intervention (week 12) and at follow-up (week 24).
  Patient overall rating: excellent / good / fair / poor
Return to sports rate | This will be assessed at the end of the intervention (week 12) and at follow-up (week 24).
  Participation: return to desired sport on pre-injury level / return to desired sport but on a lower level / return to sports but not desired sport / no return to sports
Hop test | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  Self-reported pain rating on a Visual Analogue Scale (VAS) during a single leg hop test
Lower Extremity Functional Scale | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  The lower extremity functional scale (LEFS) is a valid patient-rated outcome measure for the measurement of lower extremity function.
Tampa scale for kinesiophobia (TSK) | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  The TSK is a 17-item self report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury.
Heel-raise test | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  Participants will have to perform heel raises in standing position until thay are fatigued.
Health status using the EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire.
Pain rating (VAS) during activities of daily living | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  Self-reported pain (VAS, 0-100 mm) during activities of daily living over the last seven days. A higher score indicates more pain.
Ultrasound examination to assess the structure of the Achilles tendon insertion | This will be assessed at the start (week 0), at the end of the intervention (week 12) and at follow-up (week 24).
  Anteroposterior thickness (5 mm distal from the posterosuperior calcaneal border) - Neovascularisation (modified-Öhberg scale)
Compliance | This will be assessed weekly until the end of the intervention.
  Compliance to the exercise programme and orthotics (total percentage of prescription) will be assessed using a short online questionnaire.
Pain monitoring | This will be assessed weekly until the end of the intervention.
  Numeric Pain Rating Scale (NRS, 0-10) during exercises, after exercises and in the morning will be assessed. A higher score indicates more pain.
Adverse effects | This will be assessed weekly until the end of the intervention.
  Adverse effects resulting from the intervention
Credibility/Expectations Questionnaire | This wel be assessed at the start of the intervention (week 0)
  As participants are not blinded about their assigned intervention, it is important to determine their beliefs about the treatment. With this in mind, participants will complete the Credibility/Expectations Questionnaire (CEQ) after being assigned to an intervention group.

OTHER OUTCOMES:
Ultrasound examination to assess presence of rectrocalcaneal bursitis and/or intratendinous calcifications | This will be assessed at baseline (week 0)
  Ultrasound examination of the Achilles tendon to assess associated presence of rectrocalcaneal bursitis and/or intratendinous calcifications at the Achilles tendon insertion
X-ray to assess presence of Haglund's deformity | This will be assessed at baseline (week 0)
  X-ray of the ankle to assess associated presence of Haglund's deformity

CONTACTS AND LOCATIONS:
Overall Officials: Luc Vanden Bossche, Principal Investigator — Department of Rehabilitation Sciences, Ghent University
Locations (1):
- Department of rehabilitation sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pringels L, Capelleman R, Van den Abeele A, Burssens A, Planckaert G, Wezenbeek E, Vanden Bossche L. Effectiveness of reducing tendon compression in the rehabilitation of insertional Achilles tendinopathy: a randomised clinical trial. Br J Sports Med. 2025 Apr 24;59(9):640-650. doi: 10.1136/bjsports-2024-109138. PMID 40011018

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05456620/SAP_000.pdf